CLINICAL TRIAL: NCT04627129
Title: A Single-center, Open, Single Does, Drug-drug Interaction Study to Investigate the Effects of Itraconazole on the Pharmacokinetics of Healthy Chinese Adult Subjects After Oral Administration of SHR2554 Tablets
Brief Title: A Itraconazole Effect Study of SHR2554 on Healthy Chinese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR2554-I-106
Record Dates: First submitted 2020-10-27; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR2554+Itraconazole (Experimental): SHR2554 50 mg QD on Day 1 and Day 8, Itraconazole 200 mg once daily (QD) from Study Day 4 - 12
  Interventions: Drug: SHR2554 and Itraconazole

INTERVENTIONS:
Drug: SHR2554 and Itraconazole — Single dose of oral administration of SHR2554 and Multiple dose of oral of Itraconazole Capsules

SUMMARY:
The primary objective of the study is to evaluate the effect of Itraconazole on pharmacokinetics of healthy Chinese adult subjects after oral administration of SHR2554 tablets.

The secondary objective of the study is to evaluate the safety of single dose of SHR2554 orally in healthy subjects.

DETAILED DESCRIPTION:
SHR2554 50 mg QD on Day 1 and Day 8, Itraconazole 200 mg once daily (QD) from Study Day 4 - 12

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to enter the study:

* The informed consent is signed before the trial, and the content, process and possible adverse reactions are fully understood;
* Be able to complete the study according to the requirements of the test scheme;
* Healthy male and female subjects aged 18 to 45 years (including both ends) on the date of signing informed consent;
* The subjects have a childbearing plan and are unwilling to take effective contraceptive measures 2 weeks before the study administration (only female subjects) and 3 months after the last administration of the drug; those who are fertile and whose serum hCG test is not negative before the study medication;
* The body weight of male subjects is no less than 50 kg and that of female subjects is no less than 45 kg. Body mass index (BMI) is in the range of 19.0-26.0 kg/m2 (including the critical value).

Exclusion Criteria:

* Allergic constitution, including severe drug allergy or drug allergy history; allergic history of SHR2554 tablets, Iitraconazole or their excipients;
* People who have a history of drug and/or alcohol abuse, have a positive alcohol or drug screening test, or have a history of drug abuse in the past five years or have used drugs within 3 months before the test;
* Smoking and alcohol addicts within 3 months before the tes (drinking 14 units of alcohol per week: 1 unit = 360 ml beer,45 ml spirits, or 150 ml wine; smoking ≥ 5 cigarettes a day) and unable to prohibit smoking and alcohol during the test period;
* A clear medical history of primary diseases of important organs such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system, etc., the investigator considers not suitable for participating in this study;
* Those who have undergone any surgery within 6 months before screening;
* Hepatotoxic drugs (such as Dapsone, Erythromycin, Fluconazole, Ketoconazole, Rifampin) have been taken for a long period of time in the 6 months before screening;
* Those who have taken any clinical trial drugs within 3 months;
* Any drug that changes liver enzyme activity was taken within 28 days before taking the study drug;
* Any prescription or over-the-counter drugs、vitamin products, health products or Chinese herbal medicine taken within 14 days before taking the study drug;
* Ingested grapefruit or products containing grapefruit, food or drink containing caffeine, xanthine or alcohol within 48 hours before taking the study drug; strenuous exercise, or other factors that affect the absorption, distribution, metabolism, and excretion of the study drug;
* Patients with abnormal vital signs (systolic blood pressure < 90 mmHg or > 140 mmHg, diastolic blood pressure < 50 mmHg or > 90 mmHg; heart rate < 50 BPM or > 100 BPM) or physical examination, electrocardiogram, laboratory examination and other abnormalities have clinical significance (subject to the judgment of clinicians);
* Color Doppler echocardiography showed that left ventricular ejection fraction (LVEF) was less than 50% or QT interval corrected by friderica method in 12 lead ECG was ≥ 480msec in female subjects and ≥ 450msec in male subjects;
* HCV antibody positive, HIV antibody positive, HBsAg positive, syphilis antibody positive;
* Participated in blood donation within 3 months before taking the study drug and donate blood ≥200 mL, or received blood transfusion;
* People with a history of fainting needles and blood, have difficulty in blood collection or cannot tolerate venipuncture blood collection;
* Women during pregnancy and lactation;
* Subjects with other factors not suitable to participate in this study as considered by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 and Day 11
  Pharmacokinetics parameter of SHR2554
AUC0-t | Day 1 and Day 11
  Pharmacokinetics parameter of SHR2554
AUC0-∞ | Day 1 and Day 11
  Pharmacokinetics parameter of SHR2554: AUC0-∞

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China